CLINICAL TRIAL: NCT06342401
Title: Development and Validation fo an Exosome-Based and Machine Learning Powered Liquid Biopsy for the Detection of Early-Onset Colorectal Cancer
Brief Title: Early Onset Colorectal Cancer Detection
Acronym: ENCODE
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/ENCODE
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Adenocarcinoma; Colorectal Cancer Stage I; Colorectal Cancer Stage IV; Colorectal Cancer Stage II; Colorectal Cancer Stage III; Colorectal Neoplasms Malignant
Keywords: Early onset; Young onset; Young adult; micro-RNA; Rectal cancer; Cancer of the young; Cancer detection; Liquid biopsy
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early onset colorectal cancer (Training cohort): Colorectal cancer diagnosed before the age of 50
  Interventions: Diagnostic Test: ENCODE
- Non-disease controls (Training cohort): Individuals free from colorectal cancer, younger than 50 years of age
  Interventions: Diagnostic Test: ENCODE
- Early onset colorectal cancer (Validation cohort): Colorectal cancer diagnosed before the age of 50
  Interventions: Diagnostic Test: ENCODE
- Non-disease controls (Validation cohort): Individuals free from colorectal cancer, younger than 50 years of age
  Interventions: Diagnostic Test: ENCODE

INTERVENTIONS:
Diagnostic Test: ENCODE — A panel of microRNA, both cell-free and exosomes, whose expression level is tested from plasma samples from patients with early onset colorectal cancer and non-disease controls.
  Other Names: ENCODE (Early oNset COlorectal cancer DEtection)

SUMMARY:
Colorectal cancer (CRC) once predominantly affected older individuals, but in recent years has witnessed a progressive increase in incidence among young adults. Once rare, early-onset colorectal cancer (EOCRC, that is, a CRC diagnosed before the age of 50) now constitutes 10-15% of all newly diagnosed CRC cases and it stands as the first cause of cancer-related death in young men and the second for young women.

This study aims to detect EOCRC with a non-invasive test, using a blood-based molecular assay based on microRNA (ribonucleic acid)

DETAILED DESCRIPTION:
The rising incidence of early-onset colorectal cancer (EOCRC) is a pressing clinical issue unique to our times, and it is expected to grow with an anticipated further 90% increase in incidence by the decade's end. Challenges persist even after reducing the CRC screening age to 45: under-45s lack routine screening and compliance in the 45-50 age group remains low, partly due to invasiveness and discomfort of standard screening methods. Urgent action is warranted to develop affordable, sensitive, and feasible screening for timely detection and improved participation. A non-invasive, patient-friendly screening test, like a blood-based assay, could address these epidemiological concerns and also attract underserved populations.

This study involves the development and validation of a liquid biopsy, assessing circulating cell-free and exosomal microRNAs (cf-miRNA and exo-miRNA, respectively) for indirect sampling of tumor tissue in the bloodstream. The researchers intend to harness machine learning and bioinformatics to create an integrated panel (with both cf-miRNAs and exo-miRNAs) to enhance the inherently high sensitivity of cf-miRNAs with the distinctive specificity of exo-miRNAs. This combined approach will not only improve the performance of a diagnostic model but will also tap into the diverse tumor biology aspects of EOCRC.

The study's core goal is to develop cost-efficient, non-invasive, clinic-friendly biomarkers with high sensitivity and specificity, aiding EOCRC detection.

The researchers intend to do so in three phases:

1. To perform comprehensive small RNA-Seq from matched cf-miRNA, exo-miRNA, cancer-derived miRNA, and mucosa-derived miRNA.
2. To develop and train two miRNA detection panels (cf-miRNA and exo-miRNA, respectively) based on advanced machine-learning models and, then, combine these two using several machine-learning models to obtain a final detection biomarker.
3. To validate the findings in an independent cohort of EOCRC and controls.

In summary, this proposal promises to improve patient care and compliance, and, ultimately, reduce mortality from EOCRC.

ELIGIBILITY:
Inclusion Criteria:

* Stage I, II, III, IV colorectal cancer (TNM classification, 8th edition) diagnosed before the age of 50 (EOCRC cases)
* Received standard diagnostic and staging procedures as per local guidelines, and at least one sample was drawn before receiving any curative-intent treatment
* Colonoscopy-proven cancer-free status at the time of study inclusion (Non-disease controls)

Exclusion Criteria:

* Hereditary colorectal cancer syndromes (identified through genetic testing)
* Inflammatory bowel diseases
* Lack of written informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals younger than 50 years of age who were diagnosed with colorectal cancer before the age of 50 (cases) or were free from colorectal cancer at the time of study inclusion (controls)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  True Positive Rate: the probability of a positive test result, conditioned on the individual truly being positive

SECONDARY OUTCOMES:
Specificity | Through study completion, an average of 1 year
  True Negative Rate: the probability of a negative test result, conditioned on the individual truly being negative
Proportion of correct predictions (true positives and true negatives) among the total cases (i.e., accuracy) | Through study completion, an average of 1 year
  A measure of trueness: proportion of correct predictions (both true positives and true negatives) among the total number of cases examined

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (13):
- City of Hope Medical Center, Duarte, California, United States
- IRCCS San Raffaele, Milan, Italy
- Japan (5):
  - Kawasaki University, Kawasaki
  - Mie University, Mie
  - National Cancer Center Hospital, Tokyo
  - Tokyo Medical and Dental University, Tokyo
  - Yamagata University, Yamagata
- Spain (6):
  - Barcelona University, Barcelona
  - Colorectal Surgery, Vall d'Hebron University Hospital, Universitat Autonoma de Barcelona UAB, Barcelona
  - Surgery Department, Hospital del Mar, Barcelona, Spain, Barcelona
  - Salamanca Biomedical Research Institute, Madrid
  - University of Salamanca-SACYL-CSIC, Salamanca, Spain, Salamanca
  - University of La Laguna, San Cristóbal de La Laguna

IPD SHARING:
Plan to Share IPD: Undecided
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Patel SG, Karlitz JJ, Yen T, Lieu CH, Boland CR. The rising tide of early-onset colorectal cancer: a comprehensive review of epidemiology, clinical features, biology, risk factors, prevention, and early detection. Lancet Gastroenterol Hepatol. 2022 Mar;7(3):262-274. doi: 10.1016/S2468-1253(21)00426-X. Epub 2022 Jan 26. PMID 35090605
- [Background] Akimoto N, Ugai T, Zhong R, Hamada T, Fujiyoshi K, Giannakis M, Wu K, Cao Y, Ng K, Ogino S. Rising incidence of early-onset colorectal cancer - a call to action. Nat Rev Clin Oncol. 2021 Apr;18(4):230-243. doi: 10.1038/s41571-020-00445-1. Epub 2020 Nov 20. PMID 33219329
- [Background] Keum N, Giovannucci E. Global burden of colorectal cancer: emerging trends, risk factors and prevention strategies. Nat Rev Gastroenterol Hepatol. 2019 Dec;16(12):713-732. doi: 10.1038/s41575-019-0189-8. Epub 2019 Aug 27. PMID 31455888
- [Background] Cavestro GM, Mannucci A, Balaguer F, Hampel H, Kupfer SS, Repici A, Sartore-Bianchi A, Seppala TT, Valentini V, Boland CR, Brand RE, Buffart TE, Burke CA, Caccialanza R, Cannizzaro R, Cascinu S, Cercek A, Crosbie EJ, Danese S, Dekker E, Daca-Alvarez M, Deni F, Dominguez-Valentin M, Eng C, Goel A, Guillem JG, Houwen BBSL, Kahi C, Kalady MF, Kastrinos F, Kuhn F, Laghi L, Latchford A, Liska D, Lynch P, Malesci A, Mauri G, Meldolesi E, Moller P, Monahan KJ, Moslein G, Murphy CC, Nass K, Ng K, Oliani C, Papaleo E, Patel SG, Puzzono M, Remo A, Ricciardiello L, Ripamonti CI, Siena S, Singh SK, Stadler ZK, Stanich PP, Syngal S, Turi S, Urso ED, Valle L, Vanni VS, Vilar E, Vitellaro M, You YN, Yurgelun MB, Zuppardo RA, Stoffel EM; Associazione Italiana Familiarita Ereditarieta Tumori; Collaborative Group of the Americas on Inherited Gastrointestinal Cancer; European Hereditary Tumour Group, and the International Society for Gastrointestinal Hereditary Tumours. Delphi Initiative for Early-Onset Colorectal Cancer (DIRECt) International Management Guidelines. Clin Gastroenterol Hepatol. 2023 Mar;21(3):581-603.e33. doi: 10.1016/j.cgh.2022.12.006. Epub 2022 Dec 20. PMID 36549470
- [Background] Ullah F, Pillai AB, Omar N, Dima D, Harichand S. Early-Onset Colorectal Cancer: Current Insights. Cancers (Basel). 2023 Jun 15;15(12):3202. doi: 10.3390/cancers15123202. PMID 37370811
- [Background] Syed H, Sommovilla J, Burke CA, McGee S, Macaron C, Heald B, Lyu R, Schmit SL, Nair K, Kamath S, Krishnamurthi S, Khorana AA, Liska D. Referral, Uptake, and Outcome of Genetic Counseling and Testing in Patients With Early-Onset Colorectal Cancer. J Natl Compr Canc Netw. 2023 Nov;21(11):1156-1163.e5. doi: 10.6004/jnccn.2023.7057. PMID 37935108
- [Background] Boardman LA, Vilar E, You YN, Samadder J. AGA Clinical Practice Update on Young Adult-Onset Colorectal Cancer Diagnosis and Management: Expert Review. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2415-2424. doi: 10.1016/j.cgh.2020.05.058. Epub 2020 Jun 7. PMID 32525015
- [Background] Rogers CR, Brooks E, Curtin K, De Vera MA, Qeadan F, Rogers TN, Petersen E, Gallagher P, Pesmen C, Johnson W, Henley C, Hickman W, Newcomb E, Korous KM, Handley MA. Protocol for #iBeatCRC: a community-based intervention to increase early-onset colorectal cancer awareness using a sequential explanatory mixed-methods approach. BMJ Open. 2021 Dec 3;11(12):e048959. doi: 10.1136/bmjopen-2021-048959. PMID 34862279
- [Derived] Mannucci A, Balaguer F, Yamada Y, Nagasaka T, Toiyama Y, Okugawa Y, Marti-Gallostra M, Jimenez-Toscano M, Vidal-Tocino R, Jimenez F, Perea J, Quintero E, Boland CR, Cavestro GM, Goel A; SECOC-ENCODER Collaborators. An Exosome-Based Liquid Biopsy for the Detection of Early-Onset Colorectal Cancer: The ENCODER Multicenter Study. Gastroenterology. 2026 Feb;170(2):330-343. doi: 10.1053/j.gastro.2025.08.013. Epub 2025 Dec 9. PMID 41364052